CLINICAL TRIAL: NCT01371461
Title: Special Drug Use Investigation for PAXIL Tablet (20mg-Clinical Symptom Progression)
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 112304
Record Dates: First submitted 2011-06-09; First posted 2011-06-10 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-05

CONDITIONS: Mental Disorders
MeSH Terms: conditions — Mental Disorders | interventions — Paroxetine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients prescribed PAXIL: Patients with depression or depressed state prescribed PAXIL during study period
  Interventions: Drug: Paroxetine

INTERVENTIONS:
Drug: Paroxetine

SUMMARY:
Overall improvement, severities and changes of specific clinical symptoms were surveyed in outpatients with depression or in a depressed state to evaluate the efficacy and safety of PAXIL tablets in patients in whom the PAXIL dose was increased and those treated with a constant dose.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who is 18 years or more
* Subjects diagnosed with depression or in a depressed state

Exclusion Criteria:

* Subjects who have been treated with paroxetine prior to this investigation
* Subjects with hypersensitivity to paroxetine
* Subjects taking monoamine oxidase inhibitors (MAOIs) or within 2 weeks of stopping treatment with MAOIs
* Concomitant use in subjects taking pimozide

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects of 18 years or more diagnosed with depression or in a depressed state, who are considered appropriate to prescribe paroxetine tablet according to the prescribing information
Sampling Method: Probability Sample
Enrollment: 390 (Actual)
Dates: Start 2004-01; Primary Completion 2004-07 (Actual); Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events in Japanese subjects treated with paroxetine tablet based on prescribing information under the conditions of general clinical practice | 12 weeks
Efficacy evaluation based on Beck Depression Inventory - Second Edition (BDI-II) | 12 weeks
  The investigator asked the patient to fill out a set of self-administered BDI-II forms at each time of the patient's visits to the medical center (Patients were to make visits around 1, 2, 4, 8 and 12 weeks after starting PAXIL).
Efficacy evaluation based on overall improvement | 12 weeks
  The investigator comprehensively assessed the general condition of the patient at each time of the patient's visits to the medical center and rated the condition on a seven-grade eight-category scale (7 grades of markedly improved, moderately improved, slightly improved, unchanged, slightly worsened, worsened and severely worsened; a category of unassessable).
Efficacy evaluation based on severities of specific symptoms | 12 weeks
  The investigator rated the severities of depressed mood, anxiety, feeling irritated, hypobulia, physical symptoms and sleep disorder on a four-grade scale (none, mild, moderate and severe) based on the interview and the results of BDI-II at each time of the patient's visits to the medical center (patients were to make visits around 1, 2, 4, 8 and 12 weeks after starting PAXIL).

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline